CLINICAL TRIAL: NCT04171024
Title: Transcutaneous Diaphragm Electrical StimuLAtion in Critically Ill Patients to Prevent Diaphragm Dysfunction
Brief Title: Transcutaneous Diaphragm Electrical Stimulation in Critically Ill Patients
Acronym: TESLA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Groupe Hospitalier du Havre (Other)
Responsible Party: Principal Investigator, Clément MEDRINAL, Principal Investigator, Groupe Hospitalier du Havre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019-A00782-55
Record Dates: First submitted 2019-11-08; First posted 2019-11-20 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Critical Illness; Mechanical Ventilation; Intensive Care Unit
Keywords: Diaphragm dysfunction; Transcutaneous Electrical Stimulation; Intensive care unit; Mechanical ventilation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Group (Sham Comparator): Two channels with two electrodes each were placed above and below the right and left sides of the xiphoid process within the seventh and eighth anterior intercostal space. In addition, two channels with two electrodes each were placed on the right and left midaxillary line of the seventh and eighth anterior intercostal space.
  Transcutaneous electrical stimulation settings: Frequency (2 hertz); wave length (300 µs);
  Interventions: Device: Sham electrical stimulation
- Transcutaneous diaphragm electrical stimulation group (Experimental): Two channels with two electrodes each were placed above and below the right and left sides of the xiphoid process within the seventh and eighth anterior intercostal space. In addition, two channels with two electrodes each were placed on the right and left midaxillary line of the seventh and eighth anterior intercostal space.
  Transcutaneous electrical stimulation settings: Frequency (35 hertz); wave length (300 µs); Intensity to achieve a visual contraction
  Interventions: Device: Transcutaneous diaphragm electrical stimulation

INTERVENTIONS:
Device: Sham electrical stimulation — A non invasive sham diaphragm electrical stimulation using transcutaneous thoracic probes
  Arms: Sham Group
Device: Transcutaneous diaphragm electrical stimulation — A non invasive diaphragm electrical stimulation using transcutaneous thoracic probes
  Arms: Transcutaneous diaphragm electrical stimulation group

SUMMARY:
This study evaluates the effect of a transcutaneous electrical stimulation in critically ill patients compared to a sham electrical stimulation to decrease the incidence of diaphragm dysfunction before mechanical ventilation weaning.

ELIGIBILITY:
Inclusion Criteria:

* Patients intubated and ventilated for at least 24 h
* Patients who were expected to have at least 48h after inclusion

Exclusion Criteria:

* Patient with pacemaker
* Patient under neuro muscular blocker
* Patient post thoracic or abdominal surgery
* Patient with BMI more than 35 kg/m²
* Patient with degenerative neurological pathology
* Patient with cutaneous lesion may be interfered with probes
* Patient with chronic loss of autonomy
* Patient hospitalized more than 72 hours before ICU admission
* Patient with severe chronic obstructive pulmonary disease (FEV1 < 30%)
* Patient with decision to withhold life-sustaining treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Diaphragm Thickening fraction | Once, At the start of the spontaneous breathing trial
  Diaphragm ultrasound was conducted using a 4-12-MHz linear array transducer. Diaphragm thickness was measured at end-expiration (Tdi,ee) and end inspiration (Tdi,ei), and thickening fraction (TFdi) was calculated offline as (Tdi,ei-Tdi,ee)/Tdi,ee.

SECONDARY OUTCOMES:
Diaphragm atrophy | Once a day under mechanical ventilation, throughout the study
  Diaphragm thickeness is measured each day of the study until mechanical ventilation weaning
Inspiratory strength | Once, At the start of the spontaneous breathing trial
  Maximal inspiratory pressure is measured via an electrical manometer with unidirectional valve
Cough strength | Once, At the start of the spontaneous breathing trial
  Peak expiratory cough flow is measured with the ventilator
Proportion of patients successfully liberated from the ventilator | After 3 days of spontaneous breathing
  Extubation failure is reported when a patient present a respiratory distress and need an tracheal intubation in the 48 hours past extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Medrinal, Le Havre, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Medrinal C, Machefert M, Lamia B, Bonnevie T, Gravier FE, Hilfiker R, Prieur G, Combret Y. Transcutaneous electrical diaphragmatic stimulation in mechanically ventilated patients: a randomised study. Crit Care. 2023 Aug 30;27(1):338. doi: 10.1186/s13054-023-04597-1. PMID 37649092